CLINICAL TRIAL: NCT06694259
Title: Comparison of Anatomical and Functional Outcomes of Laser Photocoagulation and Cryopexy in Patients with Rhegmatogenous Retinal Detachment Treated with Pneumatic Retinopexy: a Randomized Clinical Trial
Brief Title: Comparison of Anatomical and Functional Outcomes of Laser Photocoagulation and Cryopexy in Patients with Rhegmatogenous Retinal Detachment Treated with Pneumatic Retinopexy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Center, Split (Other)
Responsible Party: Principal Investigator, Ivan Borjan, Ophthalmologist, Clinical Hospital Center, Split
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2181-147/01/06/LJ.Z.-23-02
Record Dates: First submitted 2024-11-15; First posted 2024-11-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Rhegmatogenous Retinal Detachment
Keywords: Rhegmatogenous retinal detachment; Pneumatic retinopexy; Transscleral cryopexy; Laser photocoagulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pneumatic retinopexy with transscleral cryopexy (Active Comparator)
  Interventions: Procedure: Pneumatic retinopexy with transscleral cryopexy
- Pneumatic retinopexy with laser photocoagulation (Active Comparator)
  Interventions: Procedure: Pneumatic retinopexy with laser photocoagulation

INTERVENTIONS:
Procedure: Pneumatic retinopexy with transscleral cryopexy — Pneumatic retinopexy with transscleral cryopexy is a procedure used to treat certain types of rhegmatogenous retinal detachments.
  Procedure steps:
  Transscleral cryopexy: in this first step, the surgeon uses a cryoprobe applied to the sclera directly over the retinal tear. The cryoprobe emits extreme cold, creating a small, localized freeze that reaches the retina and seals the tear by causing a controlled scar to form. This scar tissue holds the retina in place and prevents further fluid from passing through the tear.
  Gas bubble injection: after the cryopexy, a small gas bubble (usually sulfur hexafluoride (SF6) or perfluoropropane (C3F8)) is injected into the vitreous cavity. This bubble applies upward pressure on the retina, gently pressing it against the back wall of the eye, which aids in reattaching the retina.
  Head positioning: for several days following the procedure, the patient must keep their head in a specific position so the gas bubble remains aligned with the retinal tear.
  Arms: Pneumatic retinopexy with transscleral cryopexy
Procedure: Pneumatic retinopexy with laser photocoagulation — Pneumatic retinopexy with laser photocoagulation is a minimally invasive procedure used to repair certain types of rhegmatogenous retinal detachments.
  Procedure steps:
  Gas bubble injection: a small gas bubble, usually sulfur hexafluoride (SF6) or perfluoropropane (C3F8), is injected into the vitreous cavity which rises and applies pressure to the detached retina, pressing it back against the eye wall and helping to reapproximate the retinal layers.
  Laser photocoagulation: once the retina is positioned correctly, laser is used to create small burns around the retinal tear. This laser application causes a mild inflammatory response, creating a scar around the tear and effectively "welding" the retina to the underlying tissue. This seal prevents fluid from reaccumulating beneath the retina.
  Head positioning: following the procedure, the patient must keep their head in a specific position for several days. This positioning ensures that the gas bubble stays aligned with the retinal tear.
  Arms: Pneumatic retinopexy with laser photocoagulation

SUMMARY:
Rhegmatogenous Retinal Detachment is a pathological condition in which the inner layers of the retina separate from its outermost layer due to fluid entering between these layers through a retinal tear. Retinal detachment is one of the most urgent conditions in ophthalmology; if left untreated, it leads to severe vision loss and blindness. The only possible treatment is a surgical procedure to close the tear and reattach the separated retinal layers.

Currently, three techniques are used for surgically managing retinal detachment with a tear. You will undergo a technique called pneumatic retinopexy. In this procedure, reattachment of the retina is achieved by injecting sulfur hexafluoride gas (SF6) into the vitreous (the gel that fills the eye) about 4 millimeters from the corneal edge, using a very fine needle. The retinal tear is then closed by either freezing (cryotherapy) immediately before the gas injection or by laser photocoagulation after the gas is introduced.

The procedure will be done under local anesthesia, with the pupil first dilated using eye drops. After the procedure, a combination of antibiotics and corticosteroids will be instilled in the eye, followed by an ointment of the same combination, and the eye will be covered with a sterile dressing. You will need to maintain a specific head position, depending on the location of the retinal tear, for several days while the gas is present in the eye. This position helps the gas press against the tear, allowing it to heal. During this time, you should keep your head elevated, even at night, almost in a sitting position. Since the gas is lighter than the vitreous and rises within the eye, your head position should keep the tear positioned at 12 o'clock so the gas bubble can mechanically close it.

Proper patient selection is essential for this procedure: only patients with retinal tears limited to the upper half of the retina, with one or more tears within an hour area of the peripheral retina, are suitable for this technique. The gas does not need to be removed, as it will spontaneously reabsorb over 6-7 days. While it is in your eye, you will see it as a single bubble that will gradually shrink over 6-7 days before disappearing. If you experience severe pain on the first day, notify your surgeon, as gas expansion within the eye could cause a temporary rise in eye pressure in the first 24-48 hours.

You will need to remain in the same head position at home while the gas is present in your eye. While the gas is in place, you must not fly, as cabin pressure changes could cause the gas to expand. If you are unable to maintain the necessary position, this procedure may not be suitable for you, and an alternative technique would be needed.

This technique is less invasive than the two other surgical treatments for retinal detachment. It is performed under local anesthesia, is brief, carries fewer risks, and does not require additional follow-up procedures if the surgery is successful, which largely depends on your adherence to postoperative care.

DETAILED DESCRIPTION:
This study will include 40 patients with rhegmatogenous retinal detachment with one or more retinal breaks within two clock hours, limited to the upper half of the retina, who will be treated with pneumatic retinopexy. The patients will be thoroughly informed about the surgical procedure and the risks of potential complications. After a detailed clinical examination and the selection of suitable patients for this surgical method, the chosen patients will be randomized into two groups.

In the first group, patients will undergo transscleral cryopexy at the site of the retinal break (retrobulbar anesthesia will be given), guided by indirect ophthalmoscopy, during the same procedure. In the second group, after retinal reattachment, laser photocoagulation will be performed.

Before insufflation of the gas in the vitreous cavity, paracentesis of the anterior chamber will be performed to prevent increased intraocular pressure (0.2 mL of fluid will be withdrawn from the anterior chamber, with a 30-gauge needle). In both groups, patients will receive sulfur hexafluoride gas (SF6) in the vitreous space (0.5 mL). The gas will be injected with a 30-gauge needle, 3.5 or 4 mm from the corneal limbus (depending on the lens status: phakic/pseudophakic), at a moderate pace to avoid the formation of numerous little bubbles - a "fish eggs" phenomenon. Afterwards, evaluation of IOP will be performed by carefully evaluation of the central retinal artery for perfusion and confirmation of the light perception.

All patients will receive postoperative topical therapy with a combination of antibiotics and corticosteroids, and their head positioning will be adjusted according to the location of the retinal break(s) (positioned opposite to the retinal break for 5-8 days post-surgery, for 16 hours a day). Patients will receive appropriate hospital care and will be followed up in the retinal disease clinic postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rhegmatogenous retinal detachment with one or more tears within two clock hours, limited to the upper half of the retina

Exclusion Criteria:

* Patients with tears in the lower half of the retina
* Patients with multiple retinal tears covering more than two clock hours
* Patients with developed proliferative vitreoretinopathy
* Patients with vitreous hemorrhage
* Patients with opaque optical media due to other conditions that could obstruct a detailed fundus examination or the procedure itself
* Patients unable to follow postoperative head positioning instructions
* Patients under age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients who achieved primary retinal reattachment after undergoing pneumatic retinopexy during the 6-month follow-up period | From enrollment to the end of the 6-month follow-up period
The percentage of visual acuity improvement 6 months after the surgical procedure, assessed using the Snellen chart | From enrollment to the end of the 6-month follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Borjan, MD, Principal Investigator — Clinical Hospital Center, Split
Locations (1):
- Clinical Hospital Center, Split, Split, Croatia